CLINICAL TRIAL: NCT00004412
Title: Phase II Trial of Arginine Butyrate for Treatment of Refractory Leg Ulcers in Sickle Cell Disease or Beta Thalassemia
Brief Title: Phase II Randomized Trial:Arginine Butyrate Plus Standard Local Therapy in Patients With Refractory Sickle Cell Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susan P. Perrine (Other)
Collaborators: Boston Medical Center (Other); University of Illinois at Chicago (Other); Icahn School of Medicine at Mount Sinai (Other); University of Tennessee (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor-Investigator, Susan P. Perrine, Susan P. Perrine MD, Professor, Boston University School of Medicine, Boston University
Organization: Boston University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 199/13302; BUSM-FDR001376 (Other: Food & Drug Administration); IND 36,957 (Other: Food & Drug Administration)
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Skin Ulcers; Sickle Cell Anemia
Keywords: dermatologic disorders; genetic diseases and dysmorphic syndromes; hematologic disorders; rare disease; sickle cell anemia; skin ulcers; thalassemia major
MeSH Terms: conditions — Skin Ulcer; Anemia, Sickle Cell; Skin Diseases; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases; beta-Thalassemia | interventions — arginine butyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard local care dressing (Other): Each subject provided his/her own dressing e.g,standard local care includes cleaning, saline irrigation, dressing changes only for 8 weeks twice a week.
  Interventions: Other: Standard local care dressing
- Arginine Butyrate (Experimental): Arginine Butyrate IV plus Standard local care dressing for a total of 12 weeks. Low dose 500 mg/kg or, increased dose 750 mg/kg. First week AB given 5 days in a row, over 6 to 12hours.
  Interventions: Drug: Arginine Butyrate; Other: Standard local care dressing
- Crossover (Other): Patients are randomly assigned (following a table of random numbers prepared by a blinded statistician) between two arms of the study. Arm I is Standard local care dressing only, and Arm II is standard local care plus Arginine Butyrate (AB), the Investigational New Drug. Ulcers observed & traced weekly. Ulcer area calculated by computerized planimetry. After 12 weeks of therapy, if the ulcer size decreased by at least 25%, the AB may be continued for another 8 weeks (twice), or until the ulcer closes, plus an additional 2 weeks. The patients randomized to the Control Arm (standard local care) were given the option of crossing over to Arm II If, ulcers did not close after 8 weeks of standard local care.
  Interventions: Drug: Arginine Butyrate; Other: Standard local care dressing

INTERVENTIONS:
Drug: Arginine Butyrate — To determine if Arginine Butyrate accelerates healing of refractory leg ulcers over Standard Local Care alone.
  Arms: Arginine Butyrate; Crossover
Other: Standard local care dressing — To heal leg ulcers.

SUMMARY:
OBJECTIVES: I. Compare the efficacy of local care alone vs local care plus arginine butyrate in terms of healing rate in patients with refractory sickle cell ulcers.

II. Determine the effect of arginine butyrate therapy on tissue factors related to promotion or inhibition of wound healing in these patients.

III. Determine whether the regimen used in this study is appropriate for testing in pivotal trials.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms. Arm I: Patients receive arginine butyrate IV over 6-9 hours at night 5 days a week for 12 weeks, plus concurrent standard local therapy consisting of cleaning, saline irrigation, and dressing changes as prescribed by each patient's physician. Patients who experience progressive healing receive arginine butyrate 3-4 times a week. Arginine butyrate treatment may be discontinued and reinstated following a single 2 week medical complication.

Arm II: Patients receive standard local therapy alone for 12 weeks. Patients randomized to arm II may cross over to receive arginine butyrate if no or less than 25% healing is observed after 12 weeks.

Patients whose ulcers have closed by at least 15% per cycle may receive 2 additional 8-week cycles of arginine butyrate therapy and are followed for 2 months after healing is completed.

ELIGIBILITY:
PROTOCOL CRITERIA

INCLUSION:

--Disease Characteristics-- Significant sickle cell syndrome including Hemoglobin SS (HbSS), Hemoglobin S-beta thalassemia, and hemoglobin variants. Lower extremity or ankle ulcer (or ulcers) present for at least 6 months without healing --Patient Characteristics-- Age: 16-60 yrs Performance status: Not specified Hematopoietic: Not specified Hepatic: No hepatic compromise Transaminases no greater than 250 IU Renal: No renal compromise Creatinine no greater than 1.2 mg/mL (adults) Creatinine no greater than 0.9 mg/mL (teenagers) Other: Not pregnant Fertile patients must use effective contraception No poorly controlled seizure disorders No other secondary conditions that might inhibit immune function

* Prior/Concurrent Therapy Other: Must be treated with antibiotics prior to entry for complicating cellulitis or secondary infections

EXCLUSION :

--Prior/Concurrent Therapy-- Biologic therapy: chronic transfusion therapy Chemotherapy: prior or concurrent cancer chemotherapy concurrent butyrate derivatives Endocrine therapy: concurrent corticosteroid therapy Radiotherapy: Not specified Surgery: Not specified --Patient Characteristics-- Hepatic: hepatic compromise Transaminases greater than 250 IU Renal: renal compromise Creatinine greater than 1.2 mg/mL (adults) Creatinine greater than 0.9 mg/mL (teenagers) Other: pregnant; Fertile patients with no effective contraception Poorly controlled seizure disorders other secondary conditions that might inhibit immune function

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 1997-09; Primary Completion 2002-12 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas V. Faller, Study Chair — Boston University
Locations (4):
- United States (4):
  - University of Illinois College of Medicine, Chicago, Illinois
  - Boston University School of Medicine, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee

REFERENCES:
- [Result] McMahon L, Tamary H, Askin M, Adams-Graves P, Eberhardt RT, Sutton M, Wright EC, Castaneda SA, Faller DV, Perrine SP. A randomized phase II trial of Arginine Butyrate with standard local therapy in refractory sickle cell leg ulcers. Br J Haematol. 2010 Dec;151(5):516-24. doi: 10.1111/j.1365-2141.2010.08395.x. Epub 2010 Oct 19. PMID 20955402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study began 1998, contacted physicians at several medical centers with patients under their care for SCD with refractory leg ulcers. Electronic materials describing the study and its sponsor were transmitted to medical centers.
Groups:
- Standard Local Care Dressing: Standard local care includng cleaning, saline irrigation, dressing changes only for 8 weeks twice a week.
- Arginine Butyrate: Arginine Butyrate IV plus Standard local care dressing for a total of 12 weeks. Low dose 250 mg/kg or, increased dose 750 mg/kg. First week AB given 5 days in a row, over 8 to 12hours.
- Crossover: Patients are randomly assigned (following a table of random numbers prepared by a blinded statistician) between two arms of the study. Arm I is Allevyn Hydrophilic PU dressing (standard local care) only, and Arm II is standard local care plus Arginine Butyrate (AB), the Investigational New Drug. Ulcers observed & traced weekly. Ulcer area calculated by computerized planimetry. After 12 weeks of therapy, if the ulcer size decreased by at least 25%, the AB may be continued for another 8 weeks (twice), or until the ulcer closes, plus an additional 2 weeks. The patients randomized to the Control Arm ( standard local care) were given the option of crossing over to Arm II If, ulcers did not close after 8 weeks of standard local care.
Period: Randomized Period
Arm/Group | Standard Local Care Dressing | Arginine Butyrate | Crossover
Started | 11 | 12 | 0
Completed | 8 | 12 | 0
Not Completed | 3 | 0 | 0
Not completed — Moved to Crossover Period | 3 | 0 | 0
Period: Crossover Period
Arm/Group | Standard Local Care Dressing | Arginine Butyrate | Crossover
Started | 8 (Eight subjects were randomized to Standard of Care dressing Arm) | 12 (Twelve patients were randomized to the Arginine Butyrate plus Standard local care dressing Arm) | 3 (Three of Randomized Period's Arm I elected to move to Crossover Period's Crossover Arm.)
Completed | 8 (Eight subjects in this arm completed study without crossing over.) | 12 (Twelve subjects in this arm completed the study.) | 3 (Three subjects, from Arm I, who crossed- over to Arm II completed the study.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Local Care Dressing: Standard local care dressing including cleaning, saline irrigation, dressing changes only for 8 weeks twice a week.
- Crossover: Patients are randomly assigned (following a table of random numbers prepared by a blinded statistician) between two arms of the study. Arm I is Standard local care dressing only, and Arm II is standard local care plus Arginine Butyrate (AB), the Investigational New Drug. Ulcers observed & traced weekly. Ulcer area calculated by computerized planimetry. After 12 weeks of therapy, if the ulcer size decreased by at least 25%, the AB may be continued for another 8 weeks (twice), or until the ulcer closes, plus an additional 2 weeks. The patients randomized to the Control Arm ( standard local care) were given the option of crossing over to Arm II If, ulcers did not close after 8 weeks of standard local care.
- Total: Total of all reporting groups
Arm/Group | Standard Local Care Dressing | Arginine Butyrate | Crossover | Total
Number analyzed (Participants) | 8 | 12 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 3 | 23
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12.57478) | 33 (9.14985) | 31 (2.3094) | 32 (1.1547)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 1 | 11
  Male | 3 | 7 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 2 | 22
  Israel | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Healing Defined as a Decrease in Ulcer Area by at Least 25% of the Initial Area
Description: Treatment Arm: The AB is given as an IV infusion at 500 mg/kg over 6-9 hrs. 5 days per week for 12 weeks. After 12 weeks of therapy, if he ulcer has decreased by 25% , the AB may be continued for additional 8 weeks (twice) or, until ulcer closes plus 2 weeks, additionally.
  Ulcers photographed, traced, and ulcer areas calculated by computerized planimetry.
Time Frame: participants were followed for an average of 3 months
Population: Per protocol
Measure: Number; unit: percentage of healed ulcers
Units Other Than Participants: number of ulcers
Arm/Group | Standard Local Care Dressing | Arginine Butyrate
Number analyzed (Participants) | 11 | 12
Number analyzed (number of ulcers) | 25 | 37
percentage of healed ulcers | 24 | 78
Statistical Analysis 1: Comparison: Standard Local Care Dressing vs Arginine Butyrate; Percentage of ulcers undergoing partial and complete healing compared at 12 weeks. Mean Ulcer areas were calculated utilizing computerized planimetry, ulcer area tracings, and photography for baseline and 12 weeks and compared between the two study Arms; Test type: Superiority or Other; p = 0.05, Fisher Exact; Mean Difference (Final Values) = 0.5

2. Secondary Outcome: % Ulcers Which Completely Healed in Each Group, After 3 Months
Description: Control Arm: given option to crossover to Treatment Arm if, ulcers have not closed after 12 weeks standard local care alone.
Time Frame: two additional courses of 8 week cycles
Population: Per Protocol
Measure: Number; unit: percentage of completely healed ulcers
Units Other Than Participants: Number of ulcers
Arm/Group | Standard Local Care Dressing | Arginine Butyrate
Number analyzed (Participants) | 8 | 15
Number analyzed (Number of ulcers) | 25 | 48
percentage of completely healed ulcers | 8 | 31

ADVERSE EVENTS:
Groups:
- Standard Local Care Dressing: Standard local care including cleaning, saline irrigation, dressing changes only for 8 weeks twice a week.
Arm/Group | Standard Local Care Dressing | Arginine Butyrate
Serious Adverse Events (participants affected / at risk) | 5/11 | 9/15
Other Adverse Events (participants affected / at risk) | 1/11 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Local Care Dressing (N=11) | Arginine Butyrate (N=15)
Vaso-occlusive crisis (VOC)) (Blood and lymphatic system disorders) | 4 (13) | 7 (9)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
Clotted Portacath (Vascular disorders) | 0 (0) | 1 (1)
Chronic Limb Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Head & Eye Pain (Eye disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Bloody Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcer Infection (Infections and infestations) | 0 (0) | 1 (1)
Possible Celluitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pre-existing Osteomyelitis of Left Foot (Infections and infestations) | 0 (0) | 1 (1)
Pleural effusion and Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain , SOB (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Local Care Dressing (N=11) | Arginine Butyrate (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Decreased Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No